CLINICAL TRIAL: NCT00520975
Title: A Randomized Phase III Double-Blind Placebo-Controlled Trial of First-Line Chemotherapy and Trastuzumab With or Without Bevacizumab for Patients With HER-2/NEU Over-Expressing Metastatic Breast Cancer
Brief Title: Bevacizumab in Treating Patients With Metastatic Breast Cancer That Overexpresses HER-2/NEU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed early due to slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2009-00504; NCI-2009-00504 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1105 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH); U10CA023318 (NIH)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2016-12

CONDITIONS: Breast Carcinoma; Recurrent Breast Carcinoma; Stage IV Breast Cancer
Keywords: Trastuzumab; Bevacizumab; Metastatic Breast Cancer; HER2/NEU
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (chemotherapy and placebo) (Active Comparator): INDUCTION THERAPY: Patients receive trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22 and paclitaxel IV over 60 minutes with or without carboplatin IV over 60 minutes on days 1, 8, and 15. Patients also receive placebo IV over 30-90 minutes on day 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and placebo IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Other: Placebo; Biological: Trastuzumab
- Arm B (chemotherapy and bevacizumab) (Experimental): INDUCTION THERAPY: Patients receive trastuzumab and paclitaxel with or without carboplatin as in Arm A. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel; Biological: Trastuzumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF Humanized Monoclonal Antibody; Avastin
  Arms: Arm B (chemotherapy and bevacizumab)
Drug: Carboplatin — Given IV
  Other Names: CBDCA; JM-8; Paraplatin; NSC-241240
Drug: Paclitaxel — Given IV
  Other Names: Taxol; NSC 125973
Other: Placebo — Given IV
  Other Names: placebo therapy; sham therapy
  Arms: Arm A (chemotherapy and placebo)
Biological: Trastuzumab — Given IV
  Other Names: Anti-HER2 Monoclonal Antibody; Herceptin

SUMMARY:
This randomized phase III trial studies first-line chemotherapy and trastuzumab to compare how well they work when given with or without bevacizumab in treating patients with breast cancer that overexpresses human epidermal growth factor receptor 2 (HER-2/NEU) and has spread to other areas of the body. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as trastuzumab and bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of breast cancer by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether giving first-line chemotherapy together with trastuzumab is more effective with or without bevacizumab in treating patients with metastatic breast cancer that overexpresses HER-2/NEU.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate efficacy of the addition of bevacizumab in patients eligible for first-line trastuzumab with chemotherapy for HER-2/NEU overexpressing metastatic breast cancer, by assessing the progression-free survival (PFS) after initiation of combination therapy.

SECONDARY OBJECTIVES:

I. Evaluate response rates (RR) in patients with measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST]), when applicable.

II. Evaluate overall survival (OS).

III. Evaluate the proportion of progression-free at 6 months.

IV. Compare the toxicity of chemotherapy/trastuzumab to that of chemotherapy/ trastuzumab in combination with bevacizumab.

V. Evaluate left ventricular ejection fraction (LVEF) decline and clinical congestive heart failure (CHF).

EXPLORATORY OBJECTIVES:

I. Compare breast cancer symptoms and treatment related symptoms between patients receiving chemotherapy and trastuzumab with or without bevacizumab.

II. Evaluate whether PFS correlates with vascular endothelial growth factor (VEGF) levels in breast tumor tissue.

III. Analysis of circulating tumor cells and circulating endothelial cells (CEC).

1. Serially enumerate circulating tumor cells (CTC) and CEC in patients on study and determine whether: the number of CTC and CEC decrease in responding patients; the extent of CTC and CEC decrease is greater in the experimental arm, Arm B versus the control arm, Arm A; enumeration of CTC and CEC in responding patients correlate with progression free survival (PFS).
2. Perform an exploratory analysis of phosphorylation status of v-akt murine thymoma viral oncogene homolog (akt)-2 in circulating tumor cells.
3. Perform an exploratory analysis of reverse transcriptase (RT)-polymerase chain reaction (PCR) of CTC messenger ribonucleic acid (mRNA) to determine whether change in expression of selected downstream targets of bevacizumab therapy can serve as pharmacodynamic or surrogate markers of bevacizumab targeting and modulation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A:

INDUCTION THERAPY: Patients receive trastuzumab intravenously (IV) over 30-90 minutes on days 1, 8, 15, and 22 and paclitaxel IV over 60 minutes with or without carboplatin IV over 60 minutes on days 1, 8, and 15. Patients also receive placebo IV over 30-90 minutes on day 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and placebo IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

ARM B:

INDUCTION THERAPY: Patients receive trastuzumab and paclitaxel with or without carboplatin as in Arm A. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 10 years.

PROJECTED ACCRUAL: 489 patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer that overexpresses HER-2/NEU with evidence of metastatic disease and/or chest wall recurrence prior to randomization
* HER-2/NEU overexpression is defined as 3+ HER-2 positivity as measured by immunohistochemistry OR HER-2 gene amplification as measured by fluorescent in situ hybridization (FISH, e.g. Vysis), per American Society of Clinical Oncology guidelines

  * NOTE: representative diagnostic tissue must be submitted for central diagnostic review for confirmation of HER-2/NEU overexpression within two weeks following patient randomization
* Evaluable (measurable or non-measurable) disease is allowed if confirmed within 4 weeks prior to randomization
* Prior endocrine treatment in the adjuvant or metastatic setting is allowed, provided last dose given >= 2 weeks prior to randomization
* Radiation therapy is allowed provided last dose is given >= 3 weeks prior to randomization
* Adjuvant trastuzumab therapy for breast cancer is allowed provided last dose was given >= 12 months prior to diagnosis of recurrence
* Adjuvant or neoadjuvant taxane therapy for breast cancer is allowed provided last dose was given >= 12 months prior to diagnosis of recurrence
* Adjuvant or neoadjuvant therapy with lapatinib is allowed provided last dose is given >= 4 weeks prior to diagnosis of recurrence
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) =< 2 times upper limit of normal (ULN) (=< 5 times normal in patients with known liver involvement)
* Serum creatinine =< 1.5 mg/dL
* Urine protein: creatinine ratio =< 0.5 OR 24-hour urine protein < 1000 mg
* International normalized ratio (INR) =< 1.5 X ULN
* Partial thromboplastin time (PTT) =< 1.5 X ULN
* Multi gated acquisition scan (MUGA) scan or echocardiogram (ECHO) within 6 weeks prior to randomization with an left ventricular ejection fraction (LVEF) above the institutional lower limit of normal
* Patients must be able to understand and provide signed and dated written informed consent
* Major surgical procedure within 4 weeks prior to randomization is not allowed (except for non-operative biopsy, which would not be considered major surgery); treatment can not begin until seven (7) days after placement of a vascular access device
* Women must not be pregnant or breastfeeding; all females of childbearing potential must have a blood or urine test within 2 weeks prior to randomization to rule out pregnancy; women of childbearing potential and sexually active males must use an accepted and effective method of contraception
* Patients on full-dose anticoagulants (e.g., warfarin) with PT/INR > 1.5 may be eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * The patient has not active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Patients with a concurrent active malignancy except carcinoma in situ of the cervix or non-melanoma skin cancers (unless disease-free for at least 5 years at study entry) are not allowed

Exclusion Criteria:

* Prior chemotherapy, trastuzumab, or bevacizumab for metastatic breast cancer
* Patients who have had a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2 in the adjuvant or neo-adjuvant setting at any time
* Patients with grade 2-4 neuropathy
* Patients with a history or radiologic evidence of central nervous system (CNS) disease
* Patients have a current non-healing wound or fracture
* Patients have a hypersensitivity to paclitaxel or drugs using the vehicle Cremophor, Chinese hamster ovary cell products or other recombinant human antibodies
* Patients have a serious medical or psychiatric illness that would prevent ability to safely participate or provide informed consent
* Patients using any of the following drugs known to inhibit platelet function are not eligible: dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and cilostazol (Pletal)
* Clinically significant cardiovascular disease, including:

  * History of cerebrovascular (CVA) within 6 months
  * Uncontrolled hypertension
  * Myocardial infarction or unstable angina within 6 months
  * New York Heart Association class II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Clinically significant peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (373):
- United States (373):
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Saint Rose Hospital, Hayward, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Portneuf Medical Center, Pocatello, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - York Hospital, York Village, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Memorial Hospital at Easton - Shore Regional Cancer Center, Easton, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Capital Regional Medical Center, Jefferson City, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Orange Regional Medical Center, Middletown, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island
  - Avera Saint Luke's Hospital and Cancer Center, Aberdeen, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Mezzanotte-Sharpe J, ONeill A, Mayer IA, Arteaga CL, Yang XJ, Wagner LI, Cella D, Meropol NJ, Alpaugh RK, Saphner TJ, Swaney RE, Hoelzer KL, Gradishar WJ, Abramson VG, Sundaram PK, Jilani SZ, Perez EA, Lin NU, Jahanzeb M, Wolff AC, Sledge GW, Reid SA. A randomized phase III double-blind placebo-controlled trial of first-line chemotherapy and trastuzumab with or without bevacizumab for patients with HER2/neu-positive metastatic breast cancer: a trial of the ECOG-ACRIN Cancer Research Group (E1105). Breast Cancer Res Treat. 2024 Sep;207(2):275-282. doi: 10.1007/s10549-024-07417-4. Epub 2024 Jul 5. PMID 38967884
- See also: "Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive." — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-six patients were randomized between November 9, 2007 and October 28, 2009 when the trial closed due to slow accrual.
Groups:
- Arm A (Chemotherapy and Placebo): INDUCTION THERAPY: Patients receive trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22 and paclitaxel IV over 60 minutes with or without carboplatin IV over 60 minutes on days 1, 8, and 15. Patients also receive placebo IV over 30-90 minutes on day 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and placebo IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Placebo: Given IV
  Trastuzumab: Given IV
- Arm B (Chemotherapy and Bevacizumab): INDUCTION THERAPY: Patients receive trastuzumab and paclitaxel with or without carboplatin as in Arm A. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 1 week after the last dose of induction trastuzumab, patients receive trastuzumab IV over 30-90 minutes and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Bevacizumab: Given IV
  Carboplatin: Given IV
  Paclitaxel: Given IV
  Trastuzumab: Given IV
Period: Overall Study
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Started | 48 | 48
Treated and Reported Adverse Events Data | 47 | 45
Completed | 0 (Treatment continued until progression or intolerable toxicity.) | 0 (Treatment continued until progression or intolerable toxicity.)
Not Completed | 48 | 48
Not completed — Disease progression | 31 | 23
Not completed — Adverse Event | 7 | 10
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Other therapy | 2 | 4
Not completed — Other reasons | 4 | 2
Not completed — Not start protocol therapy | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab) | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Median (Full Range); unit: Years] | 55 [27 to 77] | 55 [33 to 76] | 55 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as time from date of randomization to first disease progression, new second breast primaries, or to death from any cause, whichever occurred first, otherwise cases were censored at date last documented to be free of progression. Disease progression was defined using the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Kaplan-Meier method was used to estimate the median PFS.
Time Frame: assessed every 3 months for patients within 2 years of registration, every 6 months for patients 3-5 years from registration and then yearly for up to10 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 48 | 48
Months | 11.1 [8.7 to 12.4] | 13.8 [10.6 to 22.5]
Statistical Analysis 1: Comparison: Arm A (Chemotherapy and Placebo) vs Arm B (Chemotherapy and Bevacizumab); Test type: Superiority or Other; p = 0.24, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.43 to 1.23]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization until death (event), or censored at last date known alive. Kaplan-Meier method was used to estimate the median OS.
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 48 | 48
Months | 49.1 [37.2 to 67.4] | 63.0 [34.4 to 72.8]
Statistical Analysis 1: Comparison: Arm A (Chemotherapy and Placebo) vs Arm B (Chemotherapy and Bevacizumab); Test type: Superiority or Other; p = 0.75, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.61 to 1.97]

3. Secondary Outcome: Proportion of Progression-free at 6 Months
Description: Disease progression was defined using the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Proportion of progression-free at 6 months was calculated using the Kaplan-Meier method.
Time Frame: assessed at baseline, at 3 and 6 months after study entry
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 48 | 48
proportion of participants | 0.826 [0.682 to 0.908] | 0.871 [0.735 to 0.939]

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by all randomized patients. Responses are evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and/or persistence of one or more non-target lesion(s).
Time Frame: assessed at baseline, every 12 weeks while on treatment, then very 3 months if patient is <2 years from study entry, every 6 months if 2-5 years from study entry, and annually if 6-10 years from study entry until disease progression
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 48 | 48
proportion of participants | 0.542 [0.392 to 0.686] | 0.604 [0.453 to 0.742]

5. Secondary Outcome: Number of Patients Experiencing Congestive Heart Failure
Description: Clinical congestive heart failure (CHF) was assessed using Left Ventricular Ejection Fraction (LVEF) and symptom information via the Cardiac Toxicity Form as well as symptom information collected via the Adverse Event Form. Clinical CHF was defined as symptomatic decline in LVEF to below the lower limit of normal (LLN) or symptomatic diastolic dysfunction.
Time Frame: assessed every 3 months while on treatment and at 3 months post treatment
Population: All patients who began protocol treatment
Measure: Number; unit: participants
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 47 | 45
participants | 1 | 4

6. Other Pre Specified Outcome: Change in Fatigue Level Between Baseline and Cycle 6 Induction
Description: Fatigue level was measured using Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue subscale. Participants indicated their level of fatigue across 13 items, each item on a 5-point Likert scale ranging from 0 (not at all) to 4(very much). Total score per patient was calculated by taking the reverse of each item (unless specified not to), taking the sum of those items, multiplying the sum by the number of items in the scale, and then dividing that number by the number of answered items. Total score ranged from 0 to 52 with higher scores representing less fatigue.
Time Frame: assessed at baseline and at cycle 6 induction prior to starting maintenance therapy
Population: All patients who reported their fatigue level using FACIT Fatigue subscale at both baseline and cycle 6 induction
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 26 | 30
scores on a scale | 2.0 [-5 to 13] | 3.0 [-2 to 16]

7. Other Pre Specified Outcome: Change in FACT/NCCN Breast Symptom Index (FBSI) Between Baseline and Cycle 6 Induction
Description: Participants indicated their level of breast symptoms across 8 items using the Functional Assessment of Cancer Therapy/National Comprehensive Cancer Network (FACT/NCCN) FBSI scale, each item on a 5-point Likert scale ranging from 0 (not at all) to 4(very much). Total score per patient, ranged from 0 to 32 with higher scores representing fewer symptoms.
Time Frame: assessed at baseline and at cycle 6 induction prior to starting maintenance therapy
Population: All patients who reported their fatigue level using FACIT Fatigue subscale at both baseline and cycle 6 induction
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 27 | 30
scores on a scale | 1 [-14 to 9] | 2 [-26 to 18]

8. Other Pre Specified Outcome: Change in Neurotoxicity Level Between Baseline and Cycle 6 Induction
Description: Participants indicated their level of neurotoxicity symptoms across 4 items using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) scale, each item on a 5-point Likert scale ranging from 0 (not at all) to 4(very much). Total score per patient ranged from 0 to 16 with higher scores representing fewer neurotoxic symptoms.
Time Frame: assessed at baseline and at cycle 6 induction prior to starting maintenance therapy
Population: All patients who reported their neurotoxicity level using FACT/GOG-Ntx scale at both baseline and cycle 6 induction
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 26 | 30
scores on a scale | 2 [-5 to 13] | 3 [-2 to 16]

9. Other Pre Specified Outcome: Change in Level of Experiencing Side Effects Between Baseline and Cycle 6 Induction
Description: Participants indicated their level of experiencing side effects across 1 item (Functional Assessment of Cancer Therapy [FACT] item G5) on a 5-point Likert scale ranging from 0 (not at all) to 4(very much). Total score per patient, ranged from 0 to 4 with a higher score representing better quality of life (QOL).
Time Frame: assessed at baseline and at cycle 6 induction prior to starting maintenance therapy
Population: All patients who reported their level of experiencing side effects using FACT item G5 at both baseline and cycle 6 induction
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 25 | 29
scores on a scale | 0 [-2 to 2] | 1 [-2 to 3]

10. Other Pre Specified Outcome: Number of Circulating Tumor Cells at Baseline
Description: Number of circulating tumor cells per 7.5mL blood were counted prior to starting protocol therapy
Time Frame: assessed at baseline prior to starting protocol therapy
Population: Patients who had blood sample drawn at baseline prior to starting protocol therapy
Measure: Median (Full Range); unit: number of cells per 7.5 mL blood
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Number analyzed (Participants) | 31 | 34
number of cells per 7.5 mL blood | 4 [0 to 126] | 2 [0 to 690]

11. Other Pre Specified Outcome: VEGF Levels in Breast Tumor by Immunohistochemistry Assay (Tumor Sample Has Not Been Analyzed Yet, no Results Could be Reported)
Description: Tissue sections from the primary or metastatic paraffin blocks were subjected to VEGF immunohistochemistry (IHC). The VEGF cytoplasmic staining intensity was evaluated semiquantitavely using a classification from 0 to 3, with 0 representing lack of staining, 1 = low staining intensity, 2 = intermediate staining intensity and 3 = strong staining intensity. The fraction of positively staining cells will be determined as well (0 = lack of staining, 1 ≤ 1% cell staining, 2 = 1 - 10% cell staining, 3 = 10 - 50% cell staining, 4 = 50 - 90% cells staining and 5 ≤ 90% cells staining) (48). Staining intensity score zero and fraction of positively staining cells of ≤ 1% (scores zero and 1) will be considered as absence of staining and therefore negative overexpression of VEGF.
Time Frame: assessed at baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle=4 weeks during Induction therapy, 1 cycle=3 weeks during Maintenance therapy) while on treatment and for 30 days after the end of treatment
Description: After discontinuation of treatment, severe (Grade ≥ 3) long term toxicity that had not been previously reported were collected via the Long term follow-up form using the following schedule: every 3 months within 2 years of registration, then every 6 months in years 2-5, annually afterward until year 10.
Arm/Group | Arm A (Chemotherapy and Placebo) | Arm B (Chemotherapy and Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 26/47 | 34/45
Other Adverse Events (participants affected / at risk) | 19/47 | 28/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Chemotherapy and Placebo) (N=47) | Arm B (Chemotherapy and Bevacizumab) (N=45)
Allergic reaction (Immune system disorders) | 1 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytes decreased (Investigations) | 0 | 2
Lymphopenia (Investigations) | 1 | 0
Neutrophils decreased (Investigations) | 8 | 9
Platelets decreased (Investigations) | 0 | 1
Cardiac troponin T (cTnT) increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 5 | 6
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 4
Cardiomyopathy, restrictive (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 5
Fever w/o neutropenia (General disorders) | 0 | 1
Weight loss (Investigations) | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3
Urinary hemorrhage NOS (Renal and urinary disorders) | 1 | 0
Infection w/ gr3-4 neut, bronchus (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, heart (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, catheter (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 1
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 2 | 3
Neuropathy-sensory (Nervous system disorders) | 3 | 5
Neurologic-other (Nervous system disorders) | 0 | 1
Chest/thoracic pain NOS (General disorders) | 0 | 1
Head/headache (Nervous system disorders) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain-other (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Irregular menses (Reproductive system and breast disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Chemotherapy and Placebo) (N=47) | Arm B (Chemotherapy and Bevacizumab) (N=45)
Allergic reaction (Immune system disorders) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 4 | 2
Leukocytes decreased (Investigations) | 3 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 6
Fatigue (General disorders) | 7 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 9
Nausea (Gastrointestinal disorders) | 4 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 5
Neuropathy-sensory (Nervous system disorders) | 7 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less